CLINICAL TRIAL: NCT02573064
Title: Impact of Treatment With Colistin on Mortality Bacteremia Multiresistant Acinetobacter Baumannii Sensitive Colistin in Patients Critical
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FCO-COL-2015-01
Record Dates: First submitted 2015-08-28; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Acinetobacter Infections
MeSH Terms: conditions — Acinetobacter Infections | interventions — Colistin; Tigecycline; Vancomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Colistin
Drug: Tigecycline
Drug: Vancomycin

SUMMARY:
The present study was designed to study the impact of empirical treatment with colistin empirical monotherapy and combined treatment with tigecycline and vancomycin on mortality of bacteremia Multiresistant Acinetobacter Baumannii . The main objective was to evaluate the efficacy of empirical treatment with colistin and combined targeted therapy. The different therapeutical interventions were administered following the routine clinical practice in the medical centre and the investigator did not assign specific interventions to the subjects of the study.

ELIGIBILITY:
Inclusion Criteria:

* Critics included patients ≥ 16 years with monomicrobial bloodstream infections by multiresistant acinetobacter baumannii to carbapenems and sensitive to colistin accompanied by systemic inflammatory response syndrome, provided they have received targeted treatment with colistin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critical patients with monomicrobial bloodstream infections due to monoclonal antibodies were studied; specific criteria were applied for analysis of empirical therapy and targeted therapy (113 patients).
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
All-cause 30-day mortality (crude). | 30 days

SECONDARY OUTCOMES:
All-cause 14 day mortality (crude). | 14 days

REFERENCES:
- [Derived] Amat T, Gutierrez-Pizarraya A, Machuca I, Gracia-Ahufinger I, Perez-Nadales E, Torre-Gimenez A, Garnacho-Montero J, Cisneros JM, Torre-Cisneros J. The combined use of tigecycline with high-dose colistin might not be associated with higher survival in critically ill patients with bacteraemia due to carbapenem-resistant Acinetobacter baumannii. Clin Microbiol Infect. 2018 Jun;24(6):630-634. doi: 10.1016/j.cmi.2017.09.016. Epub 2017 Sep 29. PMID 28970161